CLINICAL TRIAL: NCT00667940
Title: Effect of Faculty Development on Mini-CEX Score Reliability and Accuracy: A Randomized, Controlled Trial
Brief Title: Faculty Development to Improve Mini-CEX Ratings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: David A. Cook, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-002730
Record Dates: First submitted 2008-04-23; First posted 2008-04-28 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Faculty Development
Keywords: Medical education; faculty development; rater training; clinical competence; assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Workshop (Experimental): Rater training workshop: rater error training, performance dimension training, behavioral observation training, and frame of reference training using lecture, video, and facilitated discussion
  Interventions: Behavioral: Rater training workshop
- Delayed workshop (No Intervention): No specific intervention until after follow-up assessment, then receives same workshop.

INTERVENTIONS:
Behavioral: Rater training workshop — Rater training workshop: rater error training, performance dimension training, behavioral observation training, and frame of reference training using lecture, video, and facilitated discussion
  Arms: Workshop

SUMMARY:
We will conduct a faculty development workshop with intent to improve interrater reliability and rater accuracy. Outcomes will include interrater reliability, accuracy, and workshop evaluations.

DETAILED DESCRIPTION:
Hypothesis: An intervention for training faculty preceptors on the use of the mini-CEX will improve inter-rater reliability and classification accuracy.

Methods. We will develop a faculty development workshop aimed at improving the inter-rater reliability and accuracy of mini-CEX scores. To evaluate the workshop we will conduct a randomized, controlled trial. Preceptors will be randomly assigned to immediate or delayed workshop. The primary outcome will be inter-rater reliability of mini-CEX scores as preceptors rate videotaped resident-patient encounters before and four weeks after the workshop. We will also evaluate the accuracy of performance classifications. We will also collect mini-CEX ratings of actual resident-patient interactions one year preceding and one year following the workshop, and calculate interrater reliability.

Statistical methods. Inter-rater reliability will be determined using the intraclass correlation coefficient (ICC) and corresponding confidence intervals. ICC will be used to determine chance-corrected agreement (accuracy). Discrimination (differences in mean scores among scripted levels of performance) will also be evaluated as a measure of accuracy.

Scientific basis. Clinical performance assessments constitute a key element of resident education. The effect of rater training on the inter-rater reliability of mini-CEX scores is unknown. This workshop will utilize methods (rater error and field of reference training) shown to be effective in improving rater accuracy in non-medical fields.

Inclusion criteria. All internal medicine residency continuity clinic preceptors are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine residency continuity clinic preceptor at Mayo Clinic Rochester Minnesota

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-03; Primary Completion 2006-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Interrater reliability (videotaped resident-patient encounters) | April-June 2006

SECONDARY OUTCOMES:
Rater accuracy (agreement with scripted levels of performance on videotaped resident-patient encounters): percent agreement, chance-corrected agreement, mean scores | April-June 2006
Interrater reliability (actual resident-patient encounters) | March 2005 (historical) to June 2007

CONTACTS AND LOCATIONS:
Overall Officials: David A Cook, MD, MHPE, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Cook DA, Dupras DM, Beckman TJ, Thomas KG, Pankratz VS. Effect of rater training on reliability and accuracy of mini-CEX scores: a randomized, controlled trial. J Gen Intern Med. 2009 Jan;24(1):74-9. doi: 10.1007/s11606-008-0842-3. Epub 2008 Nov 11. PMID 19002533